CLINICAL TRIAL: NCT02906111
Title: Effects on Vaginal Health and Quality of Life in Postmenopausal Women Using Ultra Low Topic Estriol Before Vaginal Surgery for Pelvic Statics Disorders
Brief Title: Vaginal Estriol Before and Vaginal Surgery for Prolapse
Acronym: VSaE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Salvatore Caruso (Other)
Responsible Party: Sponsor-Investigator, Salvatore Caruso, Professor of Gynecology, Clinic of Gynecology, Policlinico Universitario, Catania
Organization: Policlinico Universitario, Catania (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MenSurgE2
Record Dates: First submitted 2016-08-24; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Genital Prolapse
Keywords: Estriol; Prolapse; Quality of life; Vaginal health; Vaginal surgery
MeSH Terms: conditions — Prolapse | interventions — Estriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group on estriol vaginal gel (Active Comparator): Drug: 1 g/daily of vaginal gel containing 50 μg of estriol (0.005%) for 3 weeks and then twice weekly for 9 weeks, for a complete cycle of treatment of 12 weeks
  Interventions: Drug: estriol; Procedure: vaginal surgery
- Control group, no estriol treatment (Active Comparator): Procedure: vaginal surgery
  Interventions: Procedure: vaginal surgery

INTERVENTIONS:
Drug: estriol — Study Group, treated with estriol
  Control Group, no drug treatment
  Both groups will undergo vaginal surgery for prolapse
  Arms: Study Group on estriol vaginal gel
Procedure: vaginal surgery — Control Group
  Other Names: vaginal surgery for prolapse

SUMMARY:
The purpose of this study is to determine whether the vaginal estriol before vaginal surgery for pelvic statics disorders is more efficacy of no estriol treatment on vaginal health and quality of life.

DETAILED DESCRIPTION:
The aim of this randomized study was to evaluate the efficacy of low concentration of vaginal estriol gel (0.005%, 50 micrograms/1 g vaginal gel) in women with pelvic statics disorders before vaginal surgical treatment (group A), assessing the vaginal dryness, dysuria, vaginal maturation index (VMI), pH and the Vaginal Health Index (VHI). Secondary, to investigate the changes of sexual function and QoL. Women without pre surgical estriol treatment constituted the control group (group B).

ELIGIBILITY:
Inclusion Criteria:

* genital dryness,
* irritation/burning/itching of vulvas or vagina
* decreased lubrication with sexual activity
* discomfort or pain with sexual activity
* decreased arousal, orgasm, desire
* dysuria.

Exclusion Criteria:

* previous surgeries for pelvic organ prolapse
* urinary incontinence
* usage of medication
* chronic medical illness
* body mass index (BMI) ≥ 35 kg/m2
* endometrial thickness equal to or greater than 4 mm
* abnormal uterine bleeding
* hormone-dependent malignancies
* history of thromboembolic disease
* liver disease
* usage of HT for less than 3 months
* usage of phytoestrogens within 1 month before the start of the study
* partner affected by sexual disorder
* conflicting with the partner

Ages: 56 Years to 63 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Vaginal Health Indexes | vaginal gel containing 50 µg of estriol, daily, for a complete cycle of treatment of 12 weeks

SECONDARY OUTCOMES:
QoL and sexual function were investigated by the Short Form 36 (SF-36) | vaginal gel containing 50 µg of estriol, daily, for a complete cycle of treatment of 12 weeks
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire short form (PISQ-12), respectively | vaginal gel containing 50 µg of estriol, daily, for a complete cycle of treatment of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cianci, Prof, Study Chair — Policlinico Catania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Caruso S, Cianci S, Amore FF, Ventura B, Bambili E, Spadola S, Cianci A. Quality of life and sexual function of naturally postmenopausal women on an ultralow-concentration estriol vaginal gel. Menopause. 2016 Jan;23(1):47-54. doi: 10.1097/GME.0000000000000485. PMID 26079974
- [Derived] Taithongchai A, Johnson EE, Ismail SI, Barron-Millar E, Kernohan A, Thakar R. Oestrogen therapy for treating pelvic organ prolapse in postmenopausal women. Cochrane Database Syst Rev. 2023 Jul 11;7(7):CD014592. doi: 10.1002/14651858.CD014592.pub2. PMID 37431855